CLINICAL TRIAL: NCT01201135
Title: The Impact of Growth Differentiating Factor (GDF) 15 in Sickle Cell Disease and Hereditary Spherocytosis
Brief Title: GDF 15 in Sickle Cell Disease and Hereditary Spherocytosis
Acronym: GDF 15
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Wolfson Medical Center (Other Government)
Responsible Party: Dr' Ghoti Hossam, hematology department on Wolfsson Medical Center
Other Study IDs: GDF-15CTIL
Record Dates: First submitted 2010-09-12; First posted 2010-09-14 (Estimated); Last update posted 2010-09-14 (Estimated); Status verified 2010-09

CONDITIONS: Patients With Thalassemia Intermedia,; Congenital Dyserythropoietic Anemia Type I
MeSH Terms: conditions — Anemia, Dyserythropoietic, Congenital

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Sickle cell disease
- hereditary spherocytosis.

SUMMARY:
Patients with thalassemia intermedia, congenital dyserythropoietic anemia type I , and sideroblastic anemia were found to express very high levels of serum GDF15, and this contributed to the inappropriate suppression of hepcidin with subsequent secondary iron overload.The aim of our present study is to asses the levels of GDF15 and hepcidin in patients with Sickle cell disease and hereditary spherocytosis

DETAILED DESCRIPTION:
The identification of the ferroportin/hepcidin axis has allowed the effect of erythroid activity on iron balance to be studied and has created the basis for better defining the erythroid regulators.

In iron-loading anemias, ineffective erythropoiesis suppresses hepcidin production, which result in dysregulating iron homeostasis. Miller and co-workers showed that release of cytokines like growth differentiation factor 15 (GDF15) during the process of ineffective erythropoiesis inhibits hepcidin production, thus defining a molecular link between ineffective erythropoiesis, suppression of hepcidin production and parenchymal iron loading.

ELIGIBILITY:
Inclusion Criteria:

* non

Exclusion Criteria:

* non

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study will contain 40 patients with Sickle cell disease and 40 patients with hereditary spherocytosis.
  After ICF (Informed Consent Form) has been signed by the patients the following laboratory tests will be taken once during the study:
  1. GDF 15( 3ml of serum) (at the laboratory of hematology at Wolfson Medical Center/Israel)
  2. Hepcidine (3ml of serum) (at the laboratory of Prof. T. Ganz, USA). The blood samples should be taken at least one week apart from blood transfusion.
  In case of infection or acute inflammation , blood samples should be taken only one week after resolution of these conditions.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2010-09; Primary Completion 2011-09 (Estimated); Study Completion 2011-09 (Estimated)

PRIMARY OUTCOMES:
GDF 15 | year

SECONDARY OUTCOMES:
Hepcidine | year

CONTACTS AND LOCATIONS:
Overall Officials: GHOTI HOSSAM, doctor, Principal Investigator — HEMATOLOGY DEPARTMENT ON WOLFSSON MEDICAL CENTER